CLINICAL TRIAL: NCT03910972
Title: A Phase I/II Study of the Safety, Immunogenicity, and Efficacy of Sm-TSP-2/Alhydrogel® With or Without AP 10-701 for Intestinal Schistosomiasis in Healthy Ugandan Adults
Brief Title: Sm-TSP-2 Schistosomiasis Vaccine in Healthy Ugandan Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: George Washington University (Other); Makerere University Walter Reed Project (Unknown)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Co-Director, Baylor College of Medicine
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-45791; TSP-18-03 (Other: Baylor College of Medicine (Sponsor))
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Schistosomiasis; Schistosoma Mansoni
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A, Group A (Sm-TSP-2/Alhydrogel 10 mcg) (Experimental): Sm-TSP-2/Alhydrogel Schistosomiasis Vaccine, delivered by IM injection on study days 0, 56, and 12; 10 mcg dose
  Interventions: Biological: Sm-TSP-2/Alhydrogel® vaccine
- Part A, Group B (Sm-TSP-2/Alhydrogel 10 mcg + AP 10-701) (Experimental): Sm-TSP-2/Alhydrogel Schistosomiasis Vaccine plus AP 10-701, delivered by IM injection on study days 0, 56, and 12; 10 mcg dose
  Interventions: Biological: Sm-TSP-2/Alhydrogel® vaccine plus AP 10-701
- Part A, Group C (Sm-TSP-2/Alhydrogel 30 mcg) (Experimental): Sm-TSP-2/Alhydrogel Schistosomiasis Vaccine, delivered by IM injection on study days 0, 56, and 12; 30 mcg dose
  Interventions: Biological: Sm-TSP-2/Alhydrogel® vaccine
- Part A, Group D (Sm-TSP-2/Alhydrogel 30 mcg + AP 10-701) (Experimental): Sm-TSP-2/Alhydrogel Schistosomiasis Vaccine plus AP 10-701, delivered by IM injection on study days 0, 56, and 12; 30 mcg dose
  Interventions: Biological: Sm-TSP-2/Alhydrogel® vaccine plus AP 10-701
- Part A, Group E (Sm-TSP-2/Alhydrogel 100 mcg) (Experimental): Sm-TSP-2/Alhydrogel Schistosomiasis Vaccine, delivered by IM injection on study days 0, 56, and 12; 100 mcg dose
  Interventions: Biological: Sm-TSP-2/Alhydrogel® vaccine
- Part A, Group F (Sm-TSP-2/Alhydrogel 100 mcg + AP 10-701) (Experimental): Sm-TSP-2/Alhydrogel Schistosomiasis Vaccine plus AP 10-701, delivered by IM injection on study days 0, 56, and 12; 100 mcg dose
  Interventions: Biological: Sm-TSP-2/Alhydrogel® vaccine plus AP 10-701
- Part A, Group G (HBV) (Active Comparator): Hepatitis B Vaccine
  Interventions: Biological: ENGERIX-B Hepatitis B Vaccine
- Part B, Group H (Sm-TSP-2/Alhydrogel +/- AP 10-701) (Experimental): Sm-TSP-2/Alhydrogel Schistosomiasis Vaccine, with or without AP 10-701, dose and formulation determined in Part A
  Interventions: Biological: Sm-TSP-2/Alhydrogel® vaccine
- Part B, Group I (HBV) (Active Comparator): Hepatitis B Vaccine
  Interventions: Biological: ENGERIX-B Hepatitis B Vaccine

INTERVENTIONS:
Biological: Sm-TSP-2/Alhydrogel® vaccine — The Sm-TSP-2/Alhydrogel® candidate vaccine contains recombinant Sm-TSP-2 adsorbed onto aluminum hydroxide gel (Alhydrogel®) and suspended in a solution containing 10mM imidazole buffer containing 2mM phosphate and 15% sucrose, with pH 7.4 ± 0.1. The final concentrations of Sm-TSP-2 and Alhydrogel® in the drug product are 0.1mg/ml and 0.8mg/ml respectively.
  Arms: Part A, Group A (Sm-TSP-2/Alhydrogel 10 mcg); Part A, Group C (Sm-TSP-2/Alhydrogel 30 mcg); Part A, Group E (Sm-TSP-2/Alhydrogel 100 mcg); Part B, Group H (Sm-TSP-2/Alhydrogel +/- AP 10-701)
Biological: Sm-TSP-2/Alhydrogel® vaccine plus AP 10-701 — The Sm-TSP-2/Alhydrogel® candidate vaccine co-administered with the immunostimulant, AP 10-701. b) AP 10-701, also known as Gluco-Pyranosylphospho-Lipid A Aqueous Formulation (GLA-AF), is a Toll-like Receptor-4 agonist. Point-of-injection formulations with this immunostimulant will be prepared immediately prior to vaccination by adding an appropriate volume of AP 10-701 to Sm-TSP-2/Alhydrogel® and withdrawing an appropriate volume to administer the desired amount of Sm-TSP-2 plus 5µg GLA-AF.
  Arms: Part A, Group B (Sm-TSP-2/Alhydrogel 10 mcg + AP 10-701); Part A, Group D (Sm-TSP-2/Alhydrogel 30 mcg + AP 10-701); Part A, Group F (Sm-TSP-2/Alhydrogel 100 mcg + AP 10-701)
Biological: ENGERIX-B Hepatitis B Vaccine — Recombinant hepatitis B vaccine containing 10 mcg recombinant hepatitis B surface antigen per dose
  Arms: Part A, Group G (HBV); Part B, Group I (HBV)

SUMMARY:
The study will recruit up to 290 healthy adult males and non-pregnant females into a two-part clinical trial of a vaccine to protect against schistosomiasis caused by infection with S. mansoni. Two formulations of the Sm-TSP-2 vaccine will be tested: one using Alhydrogel® only, and one using Alhydrogel® plus AP 10-701, each at 3 different doses of antigen: 10mcg, 30mcg, and 100mcg.

The first part of the study will be a Phase I dose-escalation safety and immunogenicity study followed by a Phase IIb trial in which a larger number of adults will be enrolled to assess the impact of the vaccine on infection with S. mansoni. The impact of the vaccine on infection with S. haematobium will also be assessed although this will be exploratory given that potential cross-protection against this species is only hypothetical at this point.

DETAILED DESCRIPTION:
The study will recruit up to 290 healthy adult males and non-pregnant females into a two-part clinical trial of a vaccine to protect against schistosomiasis caused by infection with S. mansoni. Two formulations of the Sm-TSP-2 vaccine will be tested: one using Alhydrogel® only, and one using Alhydrogel® plus AP 10-701, each at 3 different doses of antigen: 10mcg, 30mcg, and 100mcg.

The first part of the study will be a Phase I dose-escalation safety and immunogenicity study followed by a Phase IIb trial in which a larger number of adults will be enrolled to assess the impact of the vaccine on infection with S. mansoni. The impact of the vaccine on infection with S. haematobium will also be assessed although this will be exploratory given that potential cross-protection against this species is only hypothetical at this point.

Part A: double blind (within cohort), randomized, controlled, dose-escalation Phase 1b clinical trial in S. mansoni exposed adults living in the area of Kampala, Uganda. In each of 3 cohorts, subjects will be randomly assigned to 1 of 3 groups: Sm-TSP-2/Alhydrogel®, Sm-TSP-2/Alhydrogel®/AP 10-701, or the licensed Hepatitis B vaccine (up to 12 subjects per study vaccine group and 6 subjects in the Hepatitis B vaccine group). Subjects will receive three doses of the assigned vaccine delivered intramuscularly at approximately Days 0, 56, and 112.

Safety will be measured from the time of each study vaccination (Days 0, 56, 112 [Visits 2, 7, 12]) through 7 days after each study vaccination by the occurrence of solicited injection site and systemic reactogenicity events. Unsolicited non-serious adverse events (AEs) will be collected from the time of each study vaccination through approximately 28 days after each study vaccination. New-onset chronic medical conditions (including adverse events of special interest [AESI]) and serious adverse events (SAEs) will be collected from the time of the first study vaccination (Day 0 [Visit 2]) through approximately 9 months after the third study vaccination (Day 380 [Visit 19]). Clinical laboratory evaluations for safety will be performed on venous blood collected approximately 7 days after each study vaccination.

Immunogenicity testing will include IgG antibody responses to Sm-TSP-2 by a qualified indirect ELISA on serum obtained prior to each study vaccination (Days 0, 56, 112) and at time points after each vaccination.

Ninety subjects will be enrolled into 3 groups of 30. Recruitment and enrollment into the study will occur on an ongoing basis, with each group being recruited and vaccinated in sequence.

Part A of the study is a dose escalation trial in which escalation to the next dose cohort will be determined based on evaluation of pre-defined escalation criteria, which will be evaluated 7 days after all subjects in the currently active cohort have received their first dose of vaccine. Within each cohort, the assignment to Alhydrogel®, Alhydrogel®/AP 10-701, or Hepatitis B vaccine will be randomized and double-blinded (i.e., neither the subject nor the investigator will be aware of the formulation assigned). The study will proceed as follows:

1. Cohort 1, N=30 [10mcg Sm-TSP-2/Alhydrogel® (n=12) or 10mcg Sm-TSP-2/Alhydrogel®/ AP 10-701 (n=12) or Hepatitis B vaccine (n=6)]

   1. Enroll, randomize, and administer first dose of study vaccine or Hepatitis B vaccine to initial 6 subjects
   2. After initial 6 subjects have completed Visit 3, administer the first dose of study vaccine or Hepatitis B vaccine to the remaining 24 subjects
   3. Assess 7 day post dose 1 safety data for all subjects
   4. Make escalation decision
2. Cohort 2, N=30 [30mcg Sm-TSP-2/Alhydrogel® (n=12) or 30mcg Sm-TSP-2/Alhydrogel®/AP 10-701 (n=12) or Hepatitis B vaccine (n=6)]

   1. Enroll, randomize, and administer first dose of study vaccine or Hepatitis B vaccine to initial 6 subjects
   2. After initial 6 subjects have completed Visit 3, administer the first dose of study vaccine or Hepatitis B vaccine to the remaining 24 subjects
   3. Assess 7 day post dose 1 safety data for all subjects
   4. Make escalation decision
3. Cohort 3, N=30 [100mcg Sm-TSP-2/Alhydrogel® (n=12) or 100mcg Sm-TSP-2/Alhydrogel®/AP 10-701 (n=12) or Hepatitis B vaccine (n=6)]

   1. Enroll, randomize, and administer first dose of study vaccine or Hepatitis B vaccine to initial 6 subjects
   2. After initial 6 subjects have completed Visit 3, administer the first dose of study vaccine or Hepatitis B vaccine to remaining 24 subjects
   3. Assess 7 day post dose 1 safety data for all subjects
   4. Complete follow-up for all subjects
   5. Close the study

Part B: double blind, randomized, controlled, dose-escalation Phase IIb clinical trial in adults living in the area of Kampala, Uganda, who reside in S. mansoni endemic areas with greater than or equal to 25% prevalence in children aged 5-15 years of age. In this part of the study, up to 200 eligible Schistosoma-positive (by Kato Katz fecal thick smear or CAA) adult volunteers will be progressively enrolled and randomized to receive either Sm-TSP-2/Alhydrogel® (with or without AP 10-701) or the Hepatitis B comparator vaccine, in a 1:1 fashion. The dose and formulation (i.e., with or without the point-of-injection addition of AP 10-701) of Sm-TSP-2/Alhydrogel® that will be tested in this part of the study will be chosen based on the interim results of Part A of the trial after all participants have received their third dose of vaccine. All participants in Part B will be treated with praziquantel prior to receipt of the first vaccination.

Interim safety and anti-Sm-TSP-2 IgG antibody results up to and including Day 126 of Part A of the trial will be evaluated to determine the dose that will be tested in Part B.

Two hundred subjects will be enrolled in Part B. The 12 subjects in Part A who received the same dose/formulation of Sm-TSP-2/Alhydrogel® that is chosen for Part B will be offered the opportunity to transition to Part B for the remainder of their participation in the study.

Recruitment and enrollment into the study will occur on an ongoing basis, with participants being recruited, randomized and vaccinated in sequence. Within Part B, the assignment to Sm-TSP-2/Alhydrogel® or Hepatitis B vaccine will be randomized and double-blinded (i.e., neither the subject nor the investigator will be aware of the formulation assigned). Part B of the study will proceed as follows:

1. Cohort 4, N=200 [Sm-TSP-2/Alhydrogel® [dose and formulation TBD] (n=100) or Hepatitis B vaccine (n=100)]

Subjects will receive three doses of the assigned vaccine delivered intramuscularly at approximately Days 0, 56, and 112.

Safety will be measured from the time of each study vaccination (Days 0, 56, 112 [Visits 2, 7, 12]) through 7 days after each study vaccination by the occurrence of solicited injection site and systemic reactogenicity events. Unsolicited non-serious adverse events (AEs) will be collected from the time of each study vaccination through approximately 28 days after each study vaccination. New-onset chronic medical conditions (including adverse events of special interest [AESI]) and serious adverse events (SAEs) will be collected from the time of the first study vaccination (Day 0 [Visit 2]) through approximately 23 months after the third study vaccination (Day 800 [Visit 21]). Clinical laboratory evaluations for safety will be performed on venous blood collected approximately 7 days after each study vaccination.

Immunogenicity testing will include IgG antibody responses to Sm-TSP-2 by a qualified indirect ELISA on serum obtained prior to each study vaccination (Days 0, 56, 112) and at time points after each vaccination.

Efficacy will be evaluated by measuring the impact of vaccination with Sm-TSP-2/Alhydrogel® on fecal and urine Schistosoma egg counts and CAA positivity. After final vaccination, fecal and urine samples will be collected at 12 and 23 months following the final vaccination to determine rates and intensities of re-infection. The primary endpoint to determine the impact of vaccination on infection with S. mansoni will be incidence of infection as determined by a positive CAA test or Kato-Katz fecal thick smear. The impact of vaccination on infection with S. haematobium will be assessed as an exploratory endpoint, by means of urine microscopy for schistosome eggs.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study procedures.
2. Able to understand and comply with planned study procedures and be available for all study visits.
3. Male or non-pregnant female aged 18 to 45, inclusive at the time of enrollment.
4. Are in good health, as determined by vital signs (oral temperature, pulse, and blood pressure), medical history, and brief physical examination at screening.
5. Vital signs (oral temperature, pulse, and blood pressure) are all within normal protocol-defined ranges.
6. Laboratory tests (alanine aminotransferase [ALT], creatinine, white blood cell count (WBC), hemoglobin, and platelets) are all within protocol-defined reference ranges.
7. Urinalysis with no greater than trace protein and negative for glucose.
8. Female subjects of childbearing potential must agree to practice highly effective contraception for a minimum of 30 days prior to first vaccination and for 30 days after last vaccination.
9. Female subjects of childbearing potential must have a negative urine pregnancy test within 24 hours prior to study vaccination.
10. Able to correctly answer all questions on the informed consent comprehension questionnaire.

Exclusion Criteria:

1. Has the intention to become pregnant within 5 months after enrollment in this study.
2. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after their last study vaccination.
3. Has an acute illness, including a documented oral temperature of 38.0°C or greater, within 72 hours prior to vaccination.
4. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
5. Is immunosuppressed as a result of an underlying illness or treatment.
6. Using or intends to continue using oral or parenteral steroids, high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
7. Positive test for HIV infection.
8. Volunteer has had a history of alcohol or illicit drug abuse during the past 23 months.
9. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
10. History of a severe allergic reaction or anaphylaxis to known components of the study vaccines.
11. Has an acute or chronic medical condition that, in the opinion of the investigator, would render participation in this study unsafe or would interfere with the evaluation of responses.
12. History of splenectomy.
13. Is participating or plans to participate in another clinical trial with an interventional agent during the duration of the study.
14. Received any licensed live vaccine within 30 days or any licensed inactivated vaccine within 14 days prior to the first study vaccination.
15. Planned receipt of any vaccine from the first study vaccination through 28 days after the last study vaccination.
16. Has any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
17. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
18. Anti-Sm-TSP-2 IgE antibody level above ELISA reactivity threshold.

    Part A Only:
19. Positive hepatitis B surface antigen (HBsAg).
20. Positive confirmatory test for hepatitis C virus (HCV) infection.

    Part B Only:
21. Negative for Schistosoma mansoni eggs, as assessed by the Kato Katz fecal thick smear during screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: frequency of local and systemic reactogenicity events | 7 days post-vaccination
  Frequency of solicited injection site and systemic reactogenicity, graded by severity, on the day of each study vaccination through 7 days after each study vaccination.
Safety and Tolerability: frequency of unsolicited adverse events | 28 days post-vaccination
  Frequency of unsolicited adverse events, graded by severity, from the time of each study vaccination through approximately 1 month after each study vaccination.
Safety and Tolerability: frequency of vaccine-related Serious Adverse Events | 23 months
  Frequency of study vaccine-related Serious Adverse Events from the time of the first study vaccination through the final study visit.
Safety and Tolerability: frequency of clinical safety laboratory adverse events | 7 days post-vaccination
  Frequency of clinical safety laboratory adverse events measured 7 days after each vaccination
Safety and Tolerability: frequency of new-onset chronic medical conditions | 23 months
  Frequency of new-onset chronic medical conditions, including Adverse Events of Special Interest, through the final study visit
Efficacy: proportion of subjects with detectable S. mansoni eggs | 12 and 23 months
  Proportion of subjects with detectable S. mansoni eggs at 12 and 23 months in fecal samples, as determined by Kato Katz fecal thick smear.
Efficacy: mean S. mansoni eggs per gram of feces | 12 and 23 months
  Mean S. mansoni eggs per gram as determined by fecal microscopy (Kato Katz fecal thick smear) at 12 and 23 months.
Efficacy: Proportion of subjects with a positive CAA test | 12 and 23 months
  Proportion of subjects with a positive CAA test at 12 and 23 months.

SECONDARY OUTCOMES:
Immunogenicity: peak anti-Sm-TSP-2 IgG level | Day 126
  IgG level by qualified indirect ELISA on approximately Day 126
Immunogenicity: anti-Sm-TSP-2 IgG levels over time | Approximately 14 days after doses one and two and at Days 200, 290, 380 (Parts A and B) after final dose, and at Days 548, and 800 (Part B) after final dose.
  IgG antibody response measured by qualified indirect ELISA

OTHER OUTCOMES:
Efficacy: CAA (Part B only) | 12 and 23 months following final vaccination
  Proportion of subjects with a positive CAA test
Efficacy: fecal Schistosomal DNA | 12 and 23 months following final vaccination
  Levels of Schistosoma DNA in fecal samples, as measured by real-time PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Kibuuka, MD, Principal Investigator — Makerere University Walter Reed Project
Locations (1):
- Makerere University Walter Reed Project, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to primary and secondary objectives will be made available within 12 months of finalization of the Clinical Study Report.
Time Frame: Within 12 months of finalization of the Clinical Study Report.